CLINICAL TRIAL: NCT02349152
Title: The Effect of Intraoperative Continuous Remifentanil Infusion on Glycemic Response and Variability in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass: A Prospective, Randomized, Open Label Clinical Trial
Brief Title: Remifentanil and Glycemic Response in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kathirvel Subramaniam (Other)
Collaborators: Mylan Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kathirvel Subramaniam, Visiting Associate Professor in Anesthesiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO14110258
Record Dates: First submitted 2015-01-13; First posted 2015-01-28 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Heart Diseases; Hyperglycemia
Keywords: Cardiopulmonary bypass; Heart surgery
MeSH Terms: conditions — Heart Diseases; Hyperglycemia | interventions — Remifentanil; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil group (Experimental): Half of subjects enrolled will be randomized to the remifentanil group
  Interventions: Drug: Remifentanil
- Fentanyl group (Active Comparator): Half of subjects enrolled will be randomized to the fentanyl group
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Remifentanil — Subjects in the experimental group will receive remifentanil infusion 0.1-0.4ug/kg/minute before induction of anesthesia and continued until skin closure. During cardiopulmonary bypass, remifentanil infusion will be increased to 0.5-1 ug/kg/min as hemodynamically tolerated.
  Other Names: Ultiva
  Arms: Remifentanil group
Drug: Fentanyl — Subjects in the control group will initially receive intermittent boluses of Fentanyl in the range of 50-250 ug. Additional fentanyl can be given titrated to hemodynamic parameters throughout surgery.
  Arms: Fentanyl group

SUMMARY:
This study evaluates the effect of using remifentanil during cardiopulmonary bypass surgery to supress the hyperglycemic response in perioperative period. Half of the participants will receive continuous intravenous remifentanil during surgery, while the other half will receive intermittent intravenous fentanyl during surgery. Intermittent intravenous fentanyl administration is this institution's standard of care.

DETAILED DESCRIPTION:
Stress-induced hyperglycemia is a well-known phenomena that occurs during cardiopulmonary bypass surgery. Hyperglycemia increases the incidence of major adverse events and mortality in patients undergoing cardiac surgery.

Remifentanil, an ultra-short acting opioid analgesic, has been shown to reduce the stress response to cardiopulmonary bypass when compared to intermittent fentanyl and inhalation anesthesia. This in turn, will reduce the occurence of perioperative hyperglycemia, glycemic variability and insulin requirements in patients undergoing cardiac surgery.

NOTE;

Primary Outcome changed on 06/15/2015-Change Approved by University of Pittsburgh IRB on 06/22/2015- First patient enrolled January 2016.

Primary outcome measure; Percentage of patients with two or more than two intraoperative blood glucose levels more than 180 mg% in both groups will be estimated and the difference in this parameter between the two groups will form the primary outcome measure of this study.

ELIGIBILITY:
Inclusion Criteria:

* Open cardiac surgery through sternotomy approach (coronary artery bypass, valve surgery, and any other open heart surgeries)
* Surgery with use of cardiopulmonary bypass
* Patients over 18 years of age
* Both female and male genders
* All races

Exclusion Criteria:

* Minimally invasive heart surgery through thoracotomy approach
* Patients receiving regional analgesia such as intrathecal morphine
* Patients undergoing procedures under deep hypothermic circulatory arrest
* Patients with active infections such as acute infective endocarditis
* Emergency surgery
* Patients undergoing transplantations and ventricular assist device insertion
* Patients on any mechanical circulatory support preoperatively
* Patient's refusal
* Allergy to remifentanil
* Positive pregnancy test
* Morbid obesity
* End stage liver and kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathrivel Subramaniam, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doenst T, Wijeysundera D, Karkouti K, Zechner C, Maganti M, Rao V, Borger MA. Hyperglycemia during cardiopulmonary bypass is an independent risk factor for mortality in patients undergoing cardiac surgery. J Thorac Cardiovasc Surg. 2005 Oct;130(4):1144. doi: 10.1016/j.jtcvs.2005.05.049. PMID 16214532
- [Background] Ihn CH, Joo JD, Choi JW, Kim DW, Jeon YS, Kim YS, Jung HS, Kwon SY. Comparison of stress hormone response, interleukin-6 and anaesthetic characteristics of two anaesthetic techniques: volatile induction and maintenance of anaesthesia using sevoflurane versus total intravenous anaesthesia using propofol and remifentanil. J Int Med Res. 2009 Nov-Dec;37(6):1760-71. doi: 10.1177/147323000903700612. PMID 20146874
- [Background] Subramaniam B, Lerner A, Novack V, Khabbaz K, Paryente-Wiesmann M, Hess P, Talmor D. Increased glycemic variability in patients with elevated preoperative HbA1C predicts adverse outcomes following coronary artery bypass grafting surgery. Anesth Analg. 2014 Feb;118(2):277-287. doi: 10.1213/ANE.0000000000000100. PMID 24445629
- [Background] Shinoda T, Murakami W, Takamichi Y, Iizuka H, Tanaka M, Kuwasako Y. Effect of remifentanil infusion rate on stress response in orthopedic surgery using a tourniquet application. BMC Anesthesiol. 2013 Jul 10;13:14. doi: 10.1186/1471-2253-13-14. eCollection 2013. PMID 23837943
- [Background] Cok OY, Ozkose Z, Pasaoglu H, Yardim S. Glucose response during craniotomy: propofol-remifentanil versus isoflurane-remifentanil. Minerva Anestesiol. 2011 Dec;77(12):1141-8. Epub 2011 May 20. PMID 21602751
- [Background] Lazar HL, McDonnell M, Chipkin SR, Furnary AP, Engelman RM, Sadhu AR, Bridges CR, Haan CK, Svedjeholm R, Taegtmeyer H, Shemin RJ; Society of Thoracic Surgeons Blood Glucose Guideline Task Force. The Society of Thoracic Surgeons practice guideline series: Blood glucose management during adult cardiac surgery. Ann Thorac Surg. 2009 Feb;87(2):663-9. doi: 10.1016/j.athoracsur.2008.11.011. No abstract available. PMID 19161815
- [Derived] Subramaniam K, Sciortino C, Ruppert K, Monroe A, Esper S, Boisen M, Marquez J, Hayanga H, Badhwar V. Remifentanil and perioperative glycaemic response in cardiac surgery: an open-label randomised trial. Br J Anaesth. 2020 Jun;124(6):684-692. doi: 10.1016/j.bja.2020.01.028. Epub 2020 Apr 2. PMID 32247539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was recruited 01-06-2016. The final subject was recruited 12-28-2016. All enrolled subjects were recruited at Presbyterian Hospital in Pittsburgh, Pennsylvania.
Pre-assignment Details: No pre-assignment necessary for enrollment
Period: Overall Study
Arm/Group | Remifentanil Group | Fentanyl Group
Started | 60 | 56
Completed | 54 | 52
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil Group | Fentanyl Group | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Continuous [Mean (Full Range); unit: years] | 70.0 [32.0 to 84.0] | 71.0 [46.0 to 86.0] | 70.5 [32.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 35 | 38 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 54 | 52 | 106

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Values (More Than One ) > 180 mg%
Description: Percentage of patients with two or more intraoperative blood glucose levels greater than 180 mg/dl. Percentage in both groups will be estimated, then the difference in this statistic will form the primary outcome measure of this study.
  (Primary Outcome changed on 06/15/2015-Change Approved by University of Pittsburgh IRB on 06/22/2015- First patient enrolled January 2016)
Time Frame: Intraoperative period
Measure: Count of Participants; unit: Participants
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
Participants | 17 | 33
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; The null hypothesis that there was no difference in the percentage of patients with two or more blood glucose values greater than 180mg/dl between the two groups. Power calculation was performed based on the assumption that continuous remifentanil infusion would reduce the percentage of patients with unacceptable blood glucose values (more than one BG>180 mg/dl) to an absolute value of 20%; Test type: Superiority — Power calculation was performed based on the assumption that continuous remifentanil infusion would reduce the percentage of patients with unacceptable blood glucose values (more than one BG>180 mg/dl) to an absolute value of 20%. Under these conditions, 52 patients per group would have 90% power to detect a significant difference (alpha= 0.05) between the groups. A total of 116 patients were recruited to allow for dropouts; p = 0.001, Chi-squared; Risk Ratio (RR) = 1.9, 95% CI 2-sided [1.3 to 3.0]

2. Secondary Outcome: Insulin Requirement
Description: Average dose of insulin (Units/ml) calculated for each group in the intraoperative period
Time Frame: Intraoperative period; Induction to end of surgery
Measure: Median (Full Range); unit: Units/ml
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
Units/ml | 2.9 [0.0 to 35.1] | 8.1 [0.0 to 46.7]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Test type: Superiority — Power calculation was performed based on the assumption that continuous remifentanil infusion would reduce the percentage of patients with unacceptable blood glucose values (more than one BG > 180 mg) to an absolute value of 20%. Under these conditions, 52 patients per group would have 90% power to detect a significant difference (alpha = .05) between the groups. A total of 116 patients were recruited to allow dropouts; p = 0.004, t-test, 2 sided

3. Secondary Outcome: Number of Blood Glucose Values > 180 mg%
Description: Blood glucose values that exceed 180 mg% will be counted
Time Frame: Intraoperative period, Induction to end of surgery
Measure: Median (Full Range); unit: number of glucose values >180mg%
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
number of glucose values >180mg% | 1.2 [0 to 7] | 2 [0 to 6]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.01, Fisher Exact

4. Secondary Outcome: Mean, Peak and Trough Intraoperative Blood Glucose (mg/dl)
Description: Blood glucose measured every hour
Time Frame: Intraoperative period; Induction to end of surgery
Measure: Median (Full Range); unit: Mg/dL
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
Mg/dL
  Mean Introperative Blood Glucose | 141 [84 to 292] | 156 [68 to 348]
  Peak Intraoperative Blood Glucose | 178 [110 to 292] | 205 [133 to 348]
  Lowest Intraoperative Blood Glucose | 117 [84 to 195] | 120 [68 to 178]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Mean Intraoperative Blood Glucose; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Remifentanil Group vs Fentanyl Group; Peak Intraoperative Blood Glucose; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0003, t-test, 2 sided
Statistical Analysis 3: Comparison: Remifentanil Group vs Fentanyl Group; Lowest Intraoperative Blood Glucose; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.98, t-test, 2 sided

5. Secondary Outcome: Postoperative Blood Glucose
Description: Mean and peak blood glucose levels postoperatively
Time Frame: From ICU Admission (After Surgery) Until 24 hours postoperatively
Measure: Median (Full Range); unit: mg/dl
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
mg/dl
  Mean Postoperative Blood Glucose | 139 [62 to 309] | 139 [70 to 270]
  Peak Postoperative Blood Glucose | 185 [136 to 309] | 175 [127 to 270]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Mean post-operative glucose; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.14, t-test, 2 sided
Statistical Analysis 2: Comparison: Remifentanil Group vs Fentanyl Group; Peak Postoperative Blood Glucose; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.25, t-test, 2 sided

6. Secondary Outcome: Total Postoperative Regular Insulin
Description: Total units of regular insulin required post-operatively
Time Frame: From ICU Admission (After Surgery) Until 24 hours postoperatively
Measure: Median (Full Range); unit: International Units
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
International Units | 28.1 [0 to 196] | 23.5 [0 to 158]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.49, t-test, 2 sided

7. Secondary Outcome: Intraoperative Pre-cardiopulmonary Bypass Hemodynamic Stability
Description: Blood pressure (systolic, diastolic and mean), Heart rate every 5 minutes from induction of anesthesia till systemic heparinization before cardiopulmonary bypass
Time Frame: induction of anesthesia till systemic heparinization before cardiopulmonary bypass
Population: Resources not available to analyze
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Stress Hormone Levels-Cortisol (µg/dl)
Description: Serum cortisol levels (measured as µg/dl) taken at: Prebypass, cardiopulmonary bypass (2 samples: at start of bypass and end of bypass), postbypass, ICU 8 hours postoperative period
Time Frame: Perioperative period (Intraoperatively and 8 hours postoperatively)
Measure: Median (Full Range); unit: µg/dl
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
µg/dl
  Serum Cortisol Prebypass | 12 [2.0 to 21.0] | 12 [3.0 to 26.0]
  Serum Cortisol 30 Minute After Start of CPB | 6.0 [1.0 to 19.0] | 24.5 [7.0 to 43.0]
  Serum Cortisol End of CPB | 5.0 [1.0 to 15.0] | 29.0 [6.0 to 52.0]
  Serum Cortisol End of Surgery | 8.5 [2.0 to 27.0] | 28.0 [7.0 to 56.0]
  Serum Cortisol Postoperative (8 Hours) | 36.0 [14.0 to 81.0] | 45.0 [8.0 to 80.0]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Prebypass; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.401, t-test, 2 sided
Statistical Analysis 2: Comparison: Remifentanil Group vs Fentanyl Group; 30 minutes after the start of CPB; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Remifentanil Group vs Fentanyl Group; End of CPB; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Remifentanil Group vs Fentanyl Group; End of Surgery; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Remifentanil Group vs Fentanyl Group; Postoperative (8 hours); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.021, t-test, 2 sided

9. Secondary Outcome: Inflammatory Mediator Levels, Interleukin-1b, Interleukin 6 and Tumor Necrosis Factor (TNF) (pg/ml)
Description: Inflammatory mediator levels, Interleukin-1b (IL-1b), Interleukin 6 (IL-6) and Tumor Necrosis Factor Alpha (TNFa) (all measured in pg/ml) taken at: Prebypass, cardiopulmonary bypass (2 samples:30 min start of bypass (CPB-30) and end of bypass (CPB-END), postbypass, ICU 8 hours postoperative period
Time Frame: Perioperative period (Intraoperatively and 8 hours postoperatively)
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
pg/ml
  IL-1b Pre-bypass | 1.2 [0.9 to 9.1] | 1.2 [1.0 to 3.1]
  IL-1b CPB-30 | 1.1 [1.0 to 6.3] | 1.1 [0.9 to 3.0]
  IL-1b CPB-END | 1.2 [0.9 to 5.7] | 1.2 [0.9 to 2.8]
  IL-1b post-bypass | 1.1 [0.9 to 7.5] | 1.3 [0.9 to 3.4]
  IL-1b 8-HR | 1.2 [0.9 to 6.1] | 1.2 [0.7 to 3.8]
  IL-6 Pre-bypass | 2.8 [1.0 to 329] | 2.6 [0.8 to 38.5]
  IL-6 CPB-30 | 7.4 [1.3 to 58.7] | 10.3 [1.8 to 148]
  IL-6 CPB-END | 77.2 [5.3 to 1499] | 78.3 [6.6 to 3478]
  IL-6 post-bypass | 136 [17.2 to 2504] | 90.9 [13.2 to 8564]
  IL-6 8HR | 93.6 [5.1 to 2473] | 92.3 [16.7 to 12128]
  TNFa-Pre-bypass | 11.7 [2.1 to 29.7] | 10.4 [3.1 to 24.6]
  TNFa CPB-30 | 14.4 [5.5 to 49.7] | 12.6 [4.1 to 26.6]
  TNFa CPB-END | 18.2 [6.0 to 51.9] | 14.8 [3.6 to 56.5]
  TNFa post-bypass | 24.0 [5.3 to 136] | 17.2 [4.5 to 52.2]
  TNFa 8HR | 15.4 [1.1 to 41.8] | 11.2 [4.5 to 44.7]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the IL-1b Pre bypass; Test type: Superiority — Under these conditions, 52 patients per group would have 90% power to detect a significant difference (alpha = .05) between the groups. A total of 116 patients were recruited to allow dropouts; p = 0.580, t-test, 2 sided
Statistical Analysis 2: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the IL-1b CPB-30; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.815, t-test, 2 sided
Statistical Analysis 3: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the CPB-END; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.715, t-test, 2 sided
Statistical Analysis 4: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the IL-1b post-bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.330, t-test, 2 sided
Statistical Analysis 5: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the IL-1b 8 HR; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.651, t-test, 2 sided
Statistical Analysis 6: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the IL-6 Pre bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.439, t-test, 2 sided
Statistical Analysis 7: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the IL-6 CPB-30; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.284, t-test, 2 sided
Statistical Analysis 8: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the CPB-END; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.779, t-test, 2 sided
Statistical Analysis 9: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the IL-6 post-bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.274, t-test, 2 sided
Statistical Analysis 10: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the IL-6 8HR; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.601, t-test, 2 sided
Statistical Analysis 11: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the TNFa Pre-bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.315, t-test, 2 sided
Statistical Analysis 12: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the TNFa CPB-30; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.062, t-test, 2 sided
Statistical Analysis 13: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the TNFa CPB-END; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.090, t-test, 2 sided
Statistical Analysis 14: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the TNFa- post-bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.004, t-test, 2 sided
Statistical Analysis 15: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the TNFa-8HR; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.074, t-test, 2 sided

10. Secondary Outcome: Stress Hormone Levels-ACTH, GH, Glucagon (pg/ml)
Description: Adreno-corticotrophic hormone (ACTH), Growth Hormone (GH) and Glucagon (measured as pg/ml) taken at: Prebypass, cardiopulmonary bypass (2 samples: 30 mins after start of bypass (CPB 30) and end of bypass (CPB END), post-bypass and ICU 8 hours postoperative period
Time Frame: Perioperative period (Intraoperatively and 8 hours postoperatively)
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
pg/ml
  ACTH pre-bypass | 7.4 [1.6 to 52.1] | 7.4 [2.1 to 36.6]
  ACTH CPB-30 | 4.4 [1.8 to 27.4] | 57.8 [2.2 to 691]
  ACTH CPB-END | 4.4 [1.8 to 382] | 30.7 [2.9 to 1167]
  ACTH post-bypass | 8.0 [1.6 to 179] | 49.1 [2.7 to 6719]
  ACTH 8-hr | 77.0 [3.0 to 1022] | 41.3 [1.8 to 3351]
  GH-Pre-bypass | 495 [3.2 to 74329] | 872 [20.0 to 14106]
  GH-CPB-30 | 826 [26.0 to 88613] | 3202 [355 to 192177]
  GH-CPB-END | 947 [16.7 to 252584] | 2545 [117 to 169125]
  GH-post-bypass | 37364 [138 to 257569] | 4461 [180 to 185442]
  GH-8HR | 3658 [217 to 213721] | 2696 [145 to 208259]
  Glucagon pre-bypass | 229 [4.6 to 2715] | 192 [5.1 to 2242]
  Glucagon CPB-30 | 259 [4.8 to 1366] | 338 [6.2 to 2635]
  Glucagon CPB-End | 401 [5.7 to 3226] | 481 [8.2 to 3979]
  Glucagon post-bypass | 315 [5.0 to 2557] | 408 [6.8 to 2691]
  Glucagon 8-HR | 570 [7.5 to 2019] | 459 [5.0 to 4002]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the ACTH Pre-bypass group; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; p = 0.740, t-test, 2 sided
Statistical Analysis 2: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the ACTH CPB-30 group; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the ACTH CPB-END; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the ACTH post-bypass; Test type: Non-Inferiority — [test comment as in outcome 9, analysis 1]; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the ACTH 8-hr; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.014, t-test, 2 sided
Statistical Analysis 6: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the GH- Pre-bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.100, t-test, 2 sided
Statistical Analysis 7: Comparison: Remifentanil Group vs Fentanyl Group; GH-CPB-30; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the GH-CPB-END; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.009, t-test, 2 sided
Statistical Analysis 9: Comparison: Remifentanil Group vs Fentanyl Group; GH-Post-bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.046, t-test, 2 sided
Statistical Analysis 10: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the GH-8-hr; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.695, t-test, 2 sided
Statistical Analysis 11: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the Glucagon Pre Bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.455, t-test, 2 sided
Statistical Analysis 12: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the Glucagon CPB-30; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.059, t-test, 2 sided
Statistical Analysis 13: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the Glucagon CPB-END; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.175, t-test, 2 sided
Statistical Analysis 14: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the Glucagon Post-bypass; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.062, t-test, 2 sided
Statistical Analysis 15: Comparison: Remifentanil Group vs Fentanyl Group; Analyzing the Glucagon 8-hr; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.261, t-test, 2 sided

11. Secondary Outcome: Society of Thoracic Surgery Patient Outcomes
Description: Postoperative outcomes collected from the Society of Thoracic Surgery (STS) database. 30 day Mortality (outcome 1) and 30 day Readmission (outcome 2) cerebral vascular accident(outcome 3), prolonged mechanical ventilation (outcome 4), renal failure (outcome 5), atrial fibrillation (outcome 6), cardiac arrest (outcome 7)
Time Frame: 30 day outcomes
Measure: Number; unit: participants
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
participants
  30 day Mortality | 1 | 6
  30 day Readmission | 3 | 10
  Cerebral Vascular Accident | 0 | 2
  Prolonged mechanical ventilation | 8 | 8
  renal failure | 3 | 3
  atrial fibrillation | 24 | 18
  cardiac arrest | 3 | 3
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; 30-day mortality; Test type: Superiority; p = 0.06, Chi-squared
Statistical Analysis 2: Comparison: Remifentanil Group vs Fentanyl Group; 30-day readmission; Test type: Superiority; p = 0.03, Chi-squared
Statistical Analysis 3: Comparison: Remifentanil Group vs Fentanyl Group; Cerebral Vascular Accident; Test type: Superiority; p = 0.24, Chi-squared
Statistical Analysis 4: Comparison: Remifentanil Group vs Fentanyl Group; Prolonged Mechanical Ventilation; Test type: Superiority; p = 0.93, Chi-squared
Statistical Analysis 5: Comparison: Remifentanil Group vs Fentanyl Group; Renal Failure; Test type: Superiority; p = 1, Chi-squared
Statistical Analysis 6: Comparison: Remifentanil Group vs Fentanyl Group; Atrial Fibrillation; Test type: Superiority; p = 0.10, Chi-squared
Statistical Analysis 7: Comparison: Remifentanil Group vs Fentanyl Group; cardiac arrest; Test type: Superiority; p = 1, Chi-squared

12. Secondary Outcome: Postoperative Pain
Description: Pain scores; Every day 6 hour for 48 hours postoperative period
Time Frame: Every day 6 hour for 48 hours postoperative period
Population: This is a mixed model analysis to account for missing VAS values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
score on a scale
  Hours 0-6: number analyzed (Participants) | 46 | 44
  Hours 0-6 | 6.63 (1.66) | 7.18 (2.37)
  Hrs 7-12: number analyzed (Participants) | 46 | 46
  Hrs 7-12 | 6.53 (2.23) | 6.09 (2.19)
  Hrs 13-18: number analyzed (Participants) | 48 | 48
  Hrs 13-18 | 6.59 (2.07) | 5.18 (2.76)
  Hrs 19-24: number analyzed (Participants) | 47 | 49
  Hrs 19-24 | 5.88 (2.28) | 5.73 (2.38)
  Hrs 25-30: number analyzed (Participants) | 44 | 41
  Hrs 25-30 | 5.94 (5.94) | 5.65 (2.25)
  Hrs 31-36: number analyzed (Participants) | 41 | 41
  Hrs 31-36 | 5.89 (2.31) | 5.94 (2.44)
  Hrs 37-42: number analyzed (Participants) | 39 | 35
  Hrs 37-42 | 5.57 (2.35) | 5.18 (2.70)
  Hrs 43-48: number analyzed (Participants) | 31 | 25
  Hrs 43-48 | 5.08 (2.74) | 5.10 (3.11)
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Hrs 0-6; Test type: Superiority; p = 0.205, t-test, 2 sided
Statistical Analysis 2: Comparison: Remifentanil Group vs Fentanyl Group; Hrs 7-12; Test type: Superiority; p = 0.339, t-test, 2 sided
Statistical Analysis 3: Comparison: Remifentanil Group vs Fentanyl Group; Hrs 13-18; Test type: Superiority; p = 0.006, t-test, 2 sided
Statistical Analysis 4: Comparison: Remifentanil Group vs Fentanyl Group; Hrs 19-24; Test type: Superiority; p = 0.747, t-test, 2 sided
Statistical Analysis 5: Comparison: Remifentanil Group vs Fentanyl Group; Hrs 25-30; Test type: Superiority; p = 0.568, t-test, 2 sided
Statistical Analysis 6: Comparison: Remifentanil Group vs Fentanyl Group; Hrs 31-36; Test type: Superiority; p = 0.924, t-test, 2 sided
Statistical Analysis 7: Comparison: Remifentanil Group vs Fentanyl Group; Hrs 37-42; Test type: Superiority; p = 0.501, t-test, 2 sided
Statistical Analysis 8: Comparison: Remifentanil Group vs Fentanyl Group; Hrs 43-48; Test type: Superiority; p = 0.977, t-test, 2 sided

13. Secondary Outcome: Emergence From Anesthesia
Description: Time to extubation after completion of surgery in the operating room and intensive care unit
Time Frame: Immediate postoperative period until 30 days post-operatively
Measure: Median (Full Range); unit: Hours
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
Hours | 3 [0 to 141] | 2.5 [0 to 258]

14. Secondary Outcome: Wound Hyperalgesia
Description: Von frey hair objective testing
Time Frame: 96 hours postoperatively
Measure: Mean (Standard Deviation); unit: g/mm^2
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
g/mm^2
  Preop pain threshold | 3.24 (0.94) | 3.30 (1.08)
  48 Hr pain threshold | 3.71 (1.00) | 3.83 (1.28)
  96 hr pain threshold | 3.60 (1.08) | 3.72 (1.30)

15. Secondary Outcome: Development of Chronic Pain
Description: Telephonic call Numeric pain scale; Scale is 0-10, with 10 being the highest pain.
Time Frame: 1, 3, 6 and 12 months after discharge from the hospital
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
score on a scale
  S-LANSS 1 mo | 1 [0 to 8] | 3 [0 to 8]
  S-LANSS 3 mo | 0 [0 to 8] | 0 [0 to 6]
  S-LANSS 6 mo | 0 [0 to 3] | 0 [0 to 3]
  S-LANSS 12 mo | 0 [0 to 3] | 0 [0 to 3]

16. Secondary Outcome: Glycemic Variability
Description: Coefficient of variation in blood glucose levels. Denotes how large the fluctuations in blood glucose are. Higher numbers indicate increased variation.
Time Frame: From the start of induction till 24 hours postoperatively
Measure: Mean (Full Range); unit: Percent of Mean Glucose Level
Arm/Group | Remifentanil Group | Fentanyl Group
Number analyzed (Participants) | 54 | 52
Percent of Mean Glucose Level | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.4]
Statistical Analysis 1: Comparison: Remifentanil Group vs Fentanyl Group; Test type: Superiority; p = 0.350, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Remifentanil Group | Fentanyl Group
All-Cause Mortality (participants affected / at risk) | 3/54 | 6/52
Serious Adverse Events (participants affected / at risk) | 1/54 | 5/52
Other Adverse Events (participants affected / at risk) | 28/54 | 27/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remifentanil Group (N=54) | Fentanyl Group (N=52)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Pt readmitted for pneumonia.
Pericardial effusion/tamponade (Cardiac disorders) | 0 | 1
Stroke (Nervous system disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remifentanil Group (N=54) | Fentanyl Group (N=52)
Any postoperative complication (Surgical and medical procedures) | 28 | 27 — Sepsis, neurologic events, respiratory failure, thromboembolism, renal failure, cardiac arrest, rhythm abnormalities, multi-organ failures, readmissions, mortality. All data collected from Society of Thoracic Surgery (STS) database.
Sepsis (Surgical and medical procedures) | 4 | 4
Cerebrovascular Accident (Vascular disorders) | 0 | 2
Transient Ischemic Attacks (Vascular disorders) | 1 | 0
Prolonged Mechanical Ventilation (>72 hours) (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Reintubation (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary Thromboembolism (Vascular disorders) | 0 | 0
Venous Thromboembolism (Vascular disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 3 | 3
Dialysis (Renal and urinary disorders) | 3 | 3
Rhythm Requiring Permanent Pacemaker Insertion (Surgical and medical procedures) | 2 | 0
Rhythm Requiring Permanent Pacemaker/ACID (Surgical and medical procedures) | 0 | 2 — An ACID is a Automated Implantable Cardioverter Defibrillator
Cardiac Arrest (Cardiac disorders) | 3 | 3
Multisystem Organ Failure (General disorders) | 3 | 2
Readmission within 30 days (General disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No